CLINICAL TRIAL: NCT03975439
Title: Chronic Kidney Disease and Cardiovascular Disease Risk Assessment in Yakima County
Brief Title: Chronic Kidney Disease and Cardiovascular Disease Risk Assessment
Status: Withdrawn | Type: Observational
Why Stopped: Decided to do smaller pilot study instead
Sponsor: Pacific Northwest University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mark D. Baldwin, Principal Investigator, Pacific Northwest University of Health Sciences
Other Study IDs: 2019-004
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Hypertension | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hemoglobin A1C — Finger stick hemoglobin A1C
Diagnostic Test: Urinalysis — Urinalysis by dip stick looking for urine protein level
Diagnostic Test: Whole blood creatinine level — Finger stick looking for serum creatinine as an estimate of renal function

SUMMARY:
This study will investigate chronic kidney disease (CKD) and cardiovascular disease (CVD) risk factors in a sample population of Hispanics/Latinos and Caucasians in Yakima county that are rural dwelling. This investigation is intended to provide information on the impact rural geographical location and social determinants of health (SDOH) have on CKD and CVD risk factors.

DETAILED DESCRIPTION:
Yakima County has a large hispanic farmworker population. The peak work times are between May and September. There is a growing body of research that shows the risk of agricultural workers in work environments with extreme heat.

The purpose of this pilot study is to look at incidence of non-diagnosed chronic kidney disease within Yakima County to inform future studies to examine other factors and unique bio-markers that may help in the early diagnosis of heat related injuries in agricultural workers.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 75

Exclusion Criteria:

* Active malignancy
* Currently pregnant
* End stage renal disease requiring dialysis
* Current active treatment for diabetes mellitus
* Current care by a nephrologist for chronic kidney disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults of between the ages of 18 and 75 who do not meet the exclusion criteria and wish to undergo screening for kidney disease and diabetes.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Incidence of undiagnosed chronic kidney disease in farmworkers in Yakima County, WA | At the time of screening
  Finger stick and urinalysis will be done at the time of screening

SECONDARY OUTCOMES:
Incidence of undiagnosed diabetes mellitus in farmworkers in Yakima County, WA | At the time of screening
  Finger stick will be done at the time of screening
Incidence of undiagnosed hypertension in farmworkers in Yakima, County, WA | At the time of screening
  Measurement of blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Baldwin, DO, Principal Investigator — Pacific Northwest University of Health Science

REFERENCES:
- [Background] Hebert JR, Braun KL, Kaholokula JK, Armstead CA, Burch JB, Thompson B. Considering the Role of Stress in Populations of High-Risk, Underserved Community Networks Program Centers. Prog Community Health Partnersh. 2015;9 Suppl(0):71-82. doi: 10.1353/cpr.2015.0028. PMID 26213406
- [Background] Coronado GD, Thompson B, Tejeda S, Godina R, Chen L. Sociodemographic factors and self-management practices related to type 2 diabetes among Hispanics and non-Hispanic whites in a rural setting. J Rural Health. 2007 Winter;23(1):49-54. doi: 10.1111/j.1748-0361.2006.00067.x. PMID 17300478
- [Background] Ferdinand KC, Weitzman R, Israel M, Lee J, Purkayastha D, Jaimes EA. Efficacy and safety of aliskiren-based dual and triple combination therapies in US minority patients with stage 2 hypertension. J Am Soc Hypertens. 2011 Mar-Apr;5(2):102-13. doi: 10.1016/j.jash.2011.01.006. PMID 21414565
- [Background] Kurpas D, Mroczek B, Bielska D. Rural and urban disparities in quality of life and health-related behaviors among chronically ill patients. Rural Remote Health. 2014;14(2):2485. Epub 2014 Jun 10. PMID 24916658
- [Background] Krishna S, Gillespie KN, McBride TM. Diabetes burden and access to preventive care in the rural United States. J Rural Health. 2010 Winter;26(1):3-11. doi: 10.1111/j.1748-0361.2009.00259.x. PMID 20105262
- [Background] Melvin CL, Corbie-Smith G, Kumanyika SK, Pratt CA, Nelson C, Walker ER, Ammerman A, Ayala GX, Best LG, Cherrington AL, Economos CD, Green LW, Harman J, Hooker SP, Murray DM, Perri MG, Ricketts TC; Workshop Working Group on CVD Prevention in High-Risk Rural Communities. Developing a research agenda for cardiovascular disease prevention in high-risk rural communities. Am J Public Health. 2013 Jun;103(6):1011-21. doi: 10.2105/AJPH.2012.300984. Epub 2013 Apr 18. PMID 23597371
- [Background] Shoham DA, Vupputuri S, Kaufman JS, Kshirsagar AV, Diez Roux AV, Coresh J, Heiss G. Kidney disease and the cumulative burden of life course socioeconomic conditions: the Atherosclerosis Risk in Communities (ARIC) study. Soc Sci Med. 2008 Oct;67(8):1311-20. doi: 10.1016/j.socscimed.2008.06.007. Epub 2008 Jul 28. PMID 18667261